CLINICAL TRIAL: NCT03817658
Title: A Phase II Clinical Trial of Anti-PD-1 Antibody SHR-1210 Versus Placebo as Consolidation Chemotherapy After Radical Concurrent Chemoradiotherapy in Unresectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Phase II Study of SHR-1210 vs Placebo as Consolidation Chemotherapy After Radical Concurrent Chemoradiotherapy in Locally Advanced ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Feng Wang, Doctor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210--01
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 (Experimental): SHR-1210
  Interventions: Drug: SHR-1210
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1210 — First stage：
  Concurrent chemoradiotherapy:
  Cisplatin：25-30mg/m2 ivgtt d1;Capecitabine：800mg/m2, bid d1-5，qw，5weeks；Synchronous radiotherapy：1.8-2Gy/d，5d/W，45-50Gy。 Consolidation treatment： Cisplatin： 60-75mg/m2 ivgtt d1 Capecitabine：1000mg/m2, bid d1-14，q3w 6weeks。
  Second stage:
  SHR-1210 was administered intravenously (no prophylactic use), a fixed dose of 200 mg, and 3 mg/kg for subjects with a baseline weight <50 kg. Each infusion for 30 min (not less than 20 min, no more than 60 min), once every 2 weeks, 1 cycle every 4 weeks, the cumulative longest medication period is 12 months.
  Arms: SHR-1210
Drug: Placebo — First stage：
  Concurrent chemoradiotherapy:
  Cisplatin：25-30mg/m2 ivgtt d1;Capecitabine：800mg/m2, bid d1-5，qw，5weeks；Synchronous radiotherapy：1.8-2Gy/d，5d/W，45-50Gy。 Consolidation treatment： Cisplatin： 60-75mg/m2 ivgtt d1 Capecitabine：1000mg/m2, bid d1-14，q3w 6weeks。
  Second stage:
  Placebo was administered intravenously (no prophylactic use), a fixed dose of 200 mg, and 3 mg/kg for subjects with a baseline weight <50 kg. Each infusion for 30 min (not less than 20 min, no more than 60 min), once every 2 weeks, 1 cycle every 4 weeks, the cumulative longest medication period is 12 months.
  Arms: placebo

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of SHR-1210 vs placebo as consolidation chemotherapy after radical concurrent chemoradiotherapy for unresectable locally advanced ESCC.

DETAILED DESCRIPTION:
In China, the incidence of esophageal cancer has declined in recent years, but the mortality rate has been ranked fourth. Morbidity and mortality were ranked sixth and fourth in all malignancies, respectively. Therefore, esophageal cancer has always been a major malignant tumor that threatens the health of our residents. We designed a multicenter, randomized, double-blind, open-label phase II clinical trial of anti-PD-1 antibody SHR-1210 versus placebo as consolidation chemotherapy (CCT) after radical concurrent chemoradiotherapy for unresectable locally advanced esophageal squamous cell carcinoma (ESCC).The purpose of this study is to observe and evaluate the efficacy and safety of SHR-1210 vs placebo as consolidation chemotherapy after radical concurrent chemoradiotherapy for unresectable locally advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, both men and women;
2. Histology confirmed as esophageal squamous cell carcinoma;
3. T1bN+M0, T2N0-2M0 local progress period;
4. According to RECIST 1.1, at least one measurable lesion;
5. Tissue samples shall be provided for biomarker analysis, preferably newly acquired tissues, and patients who are unable to provide newly acquired tissues may provide 5-8 pieces of 5um thick paraffin sections that are archived and preserved;
6. ECOG: 0~1;
7. Expected survival period ≥ 12 weeks;
8. The main organs function normally, that is, the following criteria are met:

(1) Blood routine examination:

1. HB≥90g/L;
2. ANC ≥ 1.5 × 109 / L;
3. PLT ≥ 80 × 109 / L; (2) Biochemical examination:

a. ALB ≥ 30g / L; b. ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN; c. TBIL ≤ 1.5ULN; d. plasma Cr ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min; 9. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%); 10. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment And must be non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period; 11. Subjects voluntarily joined the study, signed informed consent, and were well-adhered to follow-up.

Exclusion Criteria:

1. Does not meet the above inclusion criteria;
2. Those who are allergic or metabolically dying of capecitabine and cisplatin;
3. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, Hyperthyroidism; patients with vitiligo; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
4. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppressive purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used for 2 weeks prior to enrollment;
5. Radiotherapy contraindications;
6. Patients with any severe and/or uncontrolled diseases;
7. Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg); myocardial ischemia or myocardial infarction with grade I or above, arrhythmia (including QT interval ≥480ms) and grade I cardiac insufficiency;
8. Active or uncontrolled serious infections;
9. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104 copies/ml or 2000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method);
10. Urine routine indicates that urine protein ≥ ++, and confirmed 24-hour urine protein quantitation > 1.0g;
11. Imaging shows that the tumor has invaded the important perivascular circumference or that the patient is likely to invade the important blood vessels and cause fatal bleeding during the follow-up study;
12. Pregnant or lactating women;
13. Patients with other malignancies within 5 years (except for basal cell carcinoma and cervical carcinoma in situ) that have been cured;
14. Patients with a history of psychotropic substance abuse who are unable to quit or have a mental disorder;
15. Patients who have participated in other drug clinical trials within four weeks;
16. At the discretion of the investigator, there are patients with serious concomitant disease that compromises patient safety or affects the patient's completion of the study;
17. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 year
  Evaluation of anti-PD-1 antibody SHR-1210 for progression-free survival in patients with locally advanced esophageal squamous cell carcinoma who did not develop disease after concurrent chemoradiotherapy
OS | up to 2 year
  From date of randomization until the date of death from any cause

SECONDARY OUTCOMES:
ORR | up to 2 year
  Evaluation of the objective response rate of anti-PD-1 antibody SHR-1210 versus placebo in patients with locally advanced esophageal squamous cell carcinoma who had no disease progression after concurrent chemoradiotherapy(RECIST 1.1)
DOR | up to 2 year
  defined as the time from the first determination of an objective response until the first documentation of progression assessed by BIRC per RECIST v1.1 or death, whichever comes first
Health-Related Quality of Life (HRQoL) | up to 2 year
  assessment of the patient's overall health status using European Quality of Life-Core 30 Questionnaire index (EORTC QLQ-C30).
Health-Related Quality of Life (HRQoL) | up to 2 year
  assessment of the patient's overall health status using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire esophageal cancer specific module (EORTC QLQ-OES18).
Health-Related Quality of Life (HRQoL) | up to 2 year
  assessment of the patient's overall health status using the generic health state instrument European Quality of Life- 5 Dimensions (EuroQol 5D EQ-5D-5L).
The incidence and severity of adverse events (AEs) | up to 2 year
  according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China